CLINICAL TRIAL: NCT07259889
Title: A Phase I Clinical Study Evaluating the Safety and Tolerability of CEL001 Injection in the Treatment of Advanced Solid Tumors
Brief Title: Safety and Tolerability Evaluation of CEL001 Injection in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Xiling Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Xiling Biotechnology Co., Ltd
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors (Phase 1)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose group 1 (Experimental): The specification of CEL001 injection is: 20ml per bag, containing approximately 5×10^8~1 × 10^9 NK cells; Encapsulated in cryovials and stored in liquid nitrogen at -196 ° C. There was only one participant in this group. After thawing at 37 ℃, CEL001 injection was administered intravenously with 5 × 10^8 cells/person/time. Administer once via intravenous infusion at Day 1, Day 20, Day 24, and Day 28, for a total of four doses.
  Interventions: Drug: NK cell preparation
- Dose group 2 (Experimental): The specification of CEL001 injection is: 20ml per bag, containing approximately 5×10^8~1 × 10^9 NK cells; Encapsulated in cryovials and stored in liquid nitrogen at -196 ° C. There will be three or six participants in this group. After thawing at 37 ℃, CEL001 injection was administered intravenously with 2×10^9 cells/person/time. Administer once via intravenous infusion at Day 1, Day 20, Day 24, and Day 28, for a total of four doses.
  Interventions: Drug: NK cell preparation
- Dose group 3 (Experimental): The specification of CEL001 injection is: 20ml per bag, containing approximately 5×10^8~1× 10^9 NK cells; Encapsulated in cryovials and stored in liquid nitrogen at -196 ° C. There will be three or six participants in this group. After thawing at 37 ℃, CEL001 injection was administered intravenously with 5×10^9 cells/person/time. Administer once via intravenous infusion at Day 1, Day 20, Day 24, and Day 28,for a total of four doses.
  Interventions: Drug: NK cell preparation

INTERVENTIONS:
Drug: NK cell preparation — CEL001 injection
  Other Names: CEL001 injection

SUMMARY:
This study is the first human, open label, dose escalation, and expansion phase I clinical trial aimed at evaluating the safety, tolerability, preliminary efficacy, pharmacokinetic characteristics, biomarker changes, and immunogenicity of CEL001 injection in the treatment of advanced solid tumors.

DETAILED DESCRIPTION:
This study is divided into five stages: screening period, single dose period, clearing period, multiple dose period, and follow-up period. The observation period for single dose DLT is tentatively set at 14 days after administration, while the observation period for multiple dose DLT is tentatively set at 28 days after the first dose of multiple doses. The cumulative administration time from a single dose is tentatively set at no more than 1 year, and the follow-up period is tentatively set at 2 years after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to enter this study:

  1. Age ≥ 18 years old, gender not limited;
  2. ECOG physical fitness status score: 0-1 points;
  3. Subjects with advanced or metastatic tumors diagnosed by histology or cytology, who have failed* or unable to tolerate standard treatment according to CSCO guidelines or NCCN guidelines, or lack effective treatment methods;
  4. Male subjects should weigh no less than 50 kilograms, and female subjects should weigh no less than 45 kilograms;
  5. Expected survival time exceeds 3 months;
  6. There must be at least one measurable lesion, defined as measurable according to the RECIST 1.1 standard;
  7. Prior to treatment, the main organ function meets the following criteria (no blood transfusion, long-acting EPO, or long-acting G-CSF treatment received within 14 days prior to the administration of the investigational drug, which can be reduced to 7 days for short acting EPO or G-CSF):

  <!-- -->

  1. Blood routine: Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, platelets ≥ 90 × 10^9/L, hemoglobin ≥ 90 g/L or ≥ 5.6 mmol/L;
  2. Kidney: serum creatinine ≤ 1.5 x upper limit of normal range (ULN) or Ccr ≥ 50 mL/min (estimated according to the Cockcroft Gault formula);
  3. Liver: Total bilirubin ≤ 1.5 × ULN (including liver metastasis or liver cancer subjects), AST and ALT ≤ 2.5 × ULN (including liver metastasis or liver cancer subjects ≤ 5 × ULN);
  4. Coagulation: International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 × ULN, Partially Activated Thromboplastin Time (APTT) ≤ 1.5 × ULN; 8. Women should agree to take appropriate contraceptive measures (such as intrauterine devices [IUDs], birth control pills, or condoms) during the study period and within 6 months after the end of the study. They must have a negative serum pregnancy test within 7 days prior to enrollment in the study and must be non lactating subjects; Men should agree to take appropriate contraceptive measures during the study period and within 6 months after the end of the study.

     * Standard treatment failure:

       * Non small cell lung cancer: (1) Subjects with metastatic non driver gene mutations: disease progression or recurrence after at least second-line treatment (including platinum based chemotherapy); (2) Subjects with driver gene mutations such as EGFR, ROS1, ALK in tumors should have received targeted therapy for these mutations that failed, followed by at least second-line treatment (including platinum based chemotherapy) for disease progression or recurrence;
       * Small cell lung cancer: disease progression or recurrence after receiving at least second-line treatment in the past;
       * Colorectal cancer: disease progression or recurrence after at least second-line treatment in the past (standard chemotherapy regimens include fluorouracil or its derivatives, oxaliplatin, and irinotecan, Subjects with BRAF V600E mutation have used BRAF inhibitors, and subjects with MSI-H/dMMR need to have used PD-1/PD-L1 treatment);
       * Head and neck squamous cell carcinoma: disease progression or recurrence after receiving at least second-line treatment (including platinum based chemotherapy) in the past;
       * Urethral epithelial cancer: disease progression or recurrence after receiving at least second-line treatment in the past (recommended treatment regimens in guidelines include PD-1/PD-L1 therapy, platinum based chemotherapy regimen, paclitaxel based chemotherapy regimen, vediximab, and vinblastine, and subjects with FGFR2/3 mutations have already used edatinib);
       * Esophageal cancer: disease progression or recurrence after receiving at least second-line treatment (including platinum based chemotherapy) in the past;
       * Cervical cancer: disease progression or recurrence after receiving at least second-line treatment in the past (including platinum based chemotherapy, subjects who meet PD-L1 positive or TMB-H or MSI-H/dMMR criteria must have received PD-1/PD-L1 treatment);
       * Hepatocellular carcinoma: disease progression or recurrence after receiving at least second-line treatment in the past;
       * Renal cell carcinoma: disease progression or recurrence after receiving at least second-line treatment in the past;
       * For other unspecified malignant tumors, refer to the latest guidelines of CSCO or NCCN.

Exclusion Criteria:

* Subjects who meet any of the following criteria will not be eligible to enter this study:

  1. Individuals allergic to any component of CEL001 injection, including those allergic to penicillin;
  2. Have received anti-tumor treatments such as chemotherapy, radiotherapy, biotherapy, endocrine therapy, targeted therapy, immunotherapy, or participated in other clinical trials within 4 weeks or 5 known drug half lives (whichever is shorter) before the first use of the investigational drug;
  3. Have received traditional Chinese medicine or modern Chinese medicine preparations with anti-tumor indications in the instructions within 14 days before the first administration;
  4. Within the past 5 years, have had malignant tumors other than those treated in this study (excluding cured thyroid cancer, basal cell carcinoma of the skin, and cervical carcinoma in situ);
  5. The adverse reactions of previous anti-tumor treatments have not yet recovered to NCI CTCAE v5.0 grade evaluation ≤ 1 (excluding toxicity judged by researchers to have no safety risks such as hair loss);
  6. Have undergone surgical procedures within 4 weeks prior to receiving treatment or have not fully recovered from any previous invasive procedures;
  7. If there are clinical symptoms of central nervous system metastasis or meningeal metastasis, or if there is other evidence indicating that the participant's central nervous system metastasis or meningeal metastasis has not been controlled, the researcher determines that it is not suitable for inclusion;
  8. Individuals with active infection (NCI CTCAE v5.0 ≥ 2) or any other suspected infection risk assessed by researchers;
  9. Have a history of autoimmune diseases, immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
  10. Subjects with active hepatitis B or active hepatitis C;
  11. Individuals who have previously received immunotherapy;
  12. Have a history of serious cardiovascular disease, such as severe cardiac rhythm or conduction abnormalities (requiring clinical intervention for ventricular arrhythmias, grade II-III atrioventricular block, etc.), myocardial infarction, history of coronary artery bypass surgery, heart failure, New York Heart Association (NYHA) classification of grade II or above, left ventricular ejection fraction (LVEF) ≤ 50% and thrombotic findings, male QTcF>450msec or female QTcF>470msec, etc; Subjects with a history of severe cerebrovascular disease such as stroke;
  13. It is necessary to combine other anti-tumor treatments (including various radiotherapy, chemotherapy, immunotherapy, targeted therapy, traditional Chinese medicine treatment, etc.);
  14. Have a clear history of neurological or mental disorders, including epilepsy or dementia;
  15. The researchers believe that there are other reasons why the subjects are not suitable to participate in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Treatment related adverse events (AEs) and serious adverse events (SAEs) | Up to 2 years after the last administration
  The incidence and severity of treatment-related adverse events (AEs) and serious adverse events (SAEs) after CEL001 injection infusion.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 12 months after the last administration
  The objective response rate (ORR) is defined as the proportion of participants who achieve complete response (CR) and partial response (PR), which is the optimal overall response.
Duration of response (DOR) | Up to 12 months after the last administration
  Duration of response (DOR) is defined as the time interval (in months) from the first assessment of a tumor as CR or PR (confirmed response) to the first objective record of disease progression (PD) or death from any cause.
Disease control rate (DCR) | 12 months after the last administration
  The disease control rate (DCR) defines the optimal overall efficacy as the proportion of participants who achieve complete response (CR), partial response (PR), and disease stability (SD).
Progression free survival (PFS) | 12 months after the last administration
  Progression free survival (PFS) is defined as the time interval (in months) between participants receiving study treatment for the first time and experiencing disease progression or death from any cause, whichever occurs first.
Overall survival (OS) | 12 months after the last administration of the last subject
  The overall survival (OS) is defined as the time interval (in months) between the first treatment and death from any cause.

OTHER OUTCOMES:
Cytokine(including but not limited to: IL-1 β, IL-2, IL-6, IL-10, TNF - α, IFN - γ) | up to 48 Days after administration
  To assess changes in systemic cytokine levels following administration of CEL001 Injection in patients with advanced solid tumors. Concentrations of target cytokines (IL-1β, IL-2, IL-6, IL-10, TNF-α, IFN-γ) will be measured via validated multiplex immunoassay at baseline and 48 days post the first dose (or key treatment cycles). The outcome will include the concentration of each cytokine and changes from baseline, with a focus on potential cytokine release-related signals.
Absolute counts of NK cells, T cells, B cells, Th cells, and CTLs | Up to 48 Days after administration
  To assess changes in peripheral blood immune cell populations following administration of CEL001 Injection in patients with advanced solid tumors. Absolute counts of NK cells, T cells, B cells, Th cells, and CTLs will be measured via validated flow cytometry at baseline and post-treatment (end of study or early termination). The primary focus is to document the absolute count values of each cell subset and their changes from baseline.
Anti-drug antibody (ADA) | Up to 48 Days after administration
  To assess the immunogenicity of CEL001 cells in patients with advanced solid tumors by detecting treatment-induced anti-drug antibodies (ADA) against infused cells or their associated components. Serum samples will be collected at pre-specified time points: baseline (prior to cell infusion), post-infusion (Day 20), and up to 48 days post-infusion. Samples will be analyzed using a validated tiered bioanalytical assay (screening for binding ADA, confirmation of specificity, and titer determination). Outcomes include the incidence of ADA positivity, titer dynamics, and neutralizing antibody (Nab) status (if tested).
Cmax | Up to 336 hours after administration
  To determine the peak peripheral blood concentration (Cmax) of viable CEL001 cells in patients with advanced solid tumors. Peripheral blood samples will be collected at pre-specified time points up to 336 hours post-infusion and analyzed using a validated flow cytometry method to quantify viable infused cells. Cmax is defined as the highest measured concentration of viable CEL001 cells in peripheral blood during the sampling period, reported in units of cells/μL(microliter). This parameter will characterize the in vivo engraftment peak of CEL001 cells, supporting the assessment of cell survival, activation, and optimal dosing schedules for future clinical studies.
Tmax | Up to 336 hours after administration
  To determine the time to peak peripheral blood concentration (Tmax) of viable CEL001 cells in patients with advanced solid tumors. Peripheral blood samples will be collected at pre-specified time points up to 336 hours post-infusion and analyzed using a validated flow cytometry method to quantify viable infused cells. Tmax is defined as the time elapsed from the start of cell infusion to the first occurrence of the peak concentration of viable CEL001 cells in peripheral blood. This parameter will be reported in hours and used to characterize the in vivo engraftment kinetics of CEL001, supporting the assessment of cell survival, activation, and optimal dosing schedules.
AUC | Up to 336 hours after administration
  To determine the area under the peripheral blood viable cell concentration-time curve (AUC) of CEL001 cells in patients with advanced solid tumors. Peripheral blood samples will be collected at pre-specified time points up to 336 hours post-infusion and analyzed using a validated flow cytometry method to quantify viable infused cells. AUC is defined as the total in vivo exposure of viable CEL001 cells over the sampling period, with key endpoints including AUC₀-ₜ (AUC from time 0 to the last quantifiable cell concentration) and AUC₀-∞ . This parameter will be reported with units (cells/μL(microliter)·hour) and used to characterize the total systemic engraftment and survival of CEL001 cells, supporting the assessment of cell therapy efficacy, safety, and optimal dosing schedules.
t1/2 | Up to 336 hours after administration
  To determine the elimination half-life (t₁/₂) of viable CEL001 cells in patients with advanced solid tumors. Peripheral blood samples will be collected at pre-specified time points up to 336 hours post-infusion and analyzed using a validated flow cytometry method to quantify viable infused cells. t₁/₂ is defined as the time required for the concentration of viable CEL001 cells in peripheral blood to decrease by half during the elimination phase, calculated via non-compartmental model (NCA) based on the cell concentration-time data. This parameter will be reported in hours or days and used to characterize the in vivo survival kinetics of CEL001 cells, supporting the assessment of cell engraftment duration, accumulation risk, and optimal dosing intervals for subsequent clinical studies.

CONTACTS AND LOCATIONS:
Overall Officials: Li Ning, Ph.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China